CLINICAL TRIAL: NCT01375985
Title: A Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of AVI-7100 in Healthy Subjects
Brief Title: Safety Study of Single Administration Intravenous Treatment for Influenza
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was halted after enrollment of the first cohort because of lack of funding
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7100-us-101
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — radavirsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVI-7100 (Experimental): Phosphorodiamidate morpholino antisense oligomer with positive charges on selected subunits (PMOplus™)
  Interventions: Drug: AVI-7100
- Placebo (Experimental): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVI-7100 — Single intravenous administration
  Arms: AVI-7100
Drug: Placebo — Single intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and pharmacology of single administrations of AVI-7100, a candidate treatment for influenza.

DETAILED DESCRIPTION:
Influenza A, a member of the Orthomyxoviridae family, is composed of a negative-sense,single-stranded and segmented ribonucleic acid (RNA) genome. An urgent need exists for new forms of treatment for influenza A based on (a) the known propensity of this virus to undergo both continuous low-level antigenic drift and less frequent but unpredictable major antigenic shift leading to pandemic disease, (b) the clear failure of vaccination, even when strains are reasonably matched, to prevent influenza-related illness in a significant proportion of vaccine recipients, and (c) the increased frequency of resistance to approved forms of therapy for influenza (eg, the adamantane derivatives and, more recently, the NA inhibitor, oseltamivir). AVI-7100 is an experimental phosphorodiamidate morpholino antisense oligomers with positive charges on selected subunits (PMOplus™). AVI-7100 specifically targets viral messenger RNA sequences. The present study is designed to characterize the safety, tolerability and pharmacokinetics of escalating single-administration doses of AVI-7100 in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and between the ages of 18 and 50 years in good general health
* Volunteers must be willing to use barrier methods of contraception or be of non-childbearing potential
* Volunteers must be willing to undergo a urine screen for drugs of abuse

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Any clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis
* Positive test for human immunodeficiency virus, hepatitis B or hepatitis C or known history of HIV infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | 28 days

SECONDARY OUTCOMES:
Plasma drug concentration | 28 days
Urine drug concentration | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hale, MD, Principal Investigator — Covance Clinical Research Unit; Alison Heald, MD, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States